CLINICAL TRIAL: NCT04046211
Title: Safety of Inhaled Hydrogen Gas Mixtures in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, John Kheir, Associate Professor, Harvard Medical School, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IRB-P00031196
Record Dates: First submitted 2019-07-25; First posted 2019-08-06 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Healthy
MeSH Terms: interventions — Hydrogen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hydrogen exposure (Experimental): The first two patients will be exposed to 2.4% hydrogen gas in medical air via HFNC for 24 hours. The second two patients will be exposed to the same gas for 48 hours. The final 4 patients will be exposed to the same gas for 72 hours.
  Interventions: Drug: Hydrogen

INTERVENTIONS:
Drug: Hydrogen — Gas exposure for 24, 48 or 72 hours via high flow nasal cannula.

SUMMARY:
Hydrogen gas may decrease the degree or incidence of brain injury following ischemia. The purpose of this study is to determine the safety and tolerability of inhaled hydrogen gas at the dose exposures required for a clinical efficacy study in healthy adult participants. Participants will breathe a gas mixture that contains a low concentration of hydrogen gas in air through a high flow nasal cannula. Investigators will test for any changes in breathing and neurologic status, as well as lab tests during and following the exposure period.

DETAILED DESCRIPTION:
Inhaled hydrogen gas (H2) has been shown to have significant protective effects on ischemic organs. Clinical trials abroad have shown promise that treatment of patients suffering from stroke, cardiac arrest, or heart attacks may benefit from inhaling hydrogen gas during the early recovery period.

The purpose of this study is to determine the safety and tolerability of inhaled hydrogen gas at the dose exposures required for a clinical efficacy study in healthy adult volunteers.

Study design. Eight (8) healthy adult participants will be recruited from the greater Boston area for this study. Consenting participants will be admitted to the hospital and will undergo a series of screens (questionnaires, examination, tests) to ensure suitability to participate. Eligible and consenting participants will then undergo exposure to 2.4% H2 in medical air via high flow nasal cannula for either 24 (n=2), 48 (n=2) or 72 (n=4) hours. Participants will be screened for adverse effects as follows: vital signs every 8 hours, nursing assessment of symptoms (codified based on the National Cancer Institute's Common Terminology Criteria for Adverse Events, CTCAE) every 8 hours, bedside spirometry daily, mini-mental state exam daily, physician physical exam daily, and serum testing (blood count, chemistry, liver and coagulation profile, venous blood gas) following exposure period.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 35
2. Able to remain inpatient for duration of admission (24-72 hours)

Exclusion Criteria:

1. History of any chronic illness, including respiratory disorders such as asthma, chronic obstructive pulmonary disease, prior acute lung injury or acute respiratory distress syndrome;
2. Inflammatory disorders, such as lupus erythematosus, inflammatory bowel disease;
3. Heritable disorders, such as trisomy 21, cystic fibrosis;
4. Mitochondrial disorders;
5. Currently smoking cigarettes or have a history of smoking cigarettes;
6. The regular use of prescription medications (except for contraceptive medications) within 30 days of enrollment;
7. Any lifetime inpatient hospitalization for respiratory illness;
8. Pregnancy.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Each duration group will be 50% male and 50% female.
Enrollment: 8 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Adverse effects/symptoms | During inhalation exposure
  Any adverse effects will be codified according the the NCI CTCAE v5.0
Adverse effects/symptoms | 2 hours following end of exposure period
  Any adverse effects will be codified according the the NCI CTCAE v5.0
Adverse effects/symptoms | 24 hours following end of exposure period
  Any adverse effects will be codified according the the NCI CTCAE v5.0
Adverse effects/symptoms | 5 days following end of exposure period
  Any adverse effects will be codified according the the NCI CTCAE v5.0

SECONDARY OUTCOMES:
Change in mini-mental state exam | 1 hour before end of exposure period
  Numerical change in mini mental state exam
Bedside spirometry | 1 hour before end of exposure period
  FEV1
Bedside spirometry | 1 hour before end of exposure period
  Forced vital capacity

CONTACTS AND LOCATIONS:
Overall Officials: John Kheir, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
The data will be shared only with the FDA and members of the DSMB and IRB.

REFERENCES:
- [Result] Cole AR, Perry DA, Raza A, Nedder AP, Pollack E, Regan WL, van den Bosch SJ, Polizzotti BD, Yang E, Davila D, Afacan O, Warfield SK, Ou Y, Sefton B, Everett AD, Neil JJ, Lidov HGW, Mayer JE, Kheir JN. Perioperatively Inhaled Hydrogen Gas Diminishes Neurologic Injury Following Experimental Circulatory Arrest in Swine. JACC Basic Transl Sci. 2019 Mar 27;4(2):176-187. doi: 10.1016/j.jacbts.2018.11.006. eCollection 2019 Apr. PMID 31061920